CLINICAL TRIAL: NCT02456519
Title: Quality of Postoperative Recovery in Children and Young People: The Modified QoR-15 Questionnaire
Brief Title: Quality of Postoperative Recovery in Children and Young People
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15HS03
Record Dates: First submitted 2015-05-19; First posted 2015-05-28 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2015-05

CONDITIONS: Quality of Recovery
Keywords: children; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PaedQoR-15 Questionnaire: Questionnaire to be completed by all participants
  Interventions: Other: PaedQoR-15 questionnaire

INTERVENTIONS:
Other: PaedQoR-15 questionnaire — Children/ young people and one parent/ guardian will complete the questionnaire before and after general anaesthesia for surgery or diagnostic imaging.

SUMMARY:
Provision of high-quality anaesthesia is a fundamental goal of all anaesthetic services. Establishing whether this is being achieved requires validated measures of anaesthetic outcomes but few of these exist, particularly for children.

QoR-15 (quality of recovery, 15 items) is a questionnaire that has been validated in adults and assesses the quality of postoperative recovery from surgery. The investigators have developed a modified version, the PaedQoR-15, that the investigators hope is capable of performing the same task in children and young people. The principle aim of this study is to assess whether PaedQoR-15 is a valid, reliable and clinically acceptable measure of the quality of postoperative recovery in children and young people.

The investigators would also like to consider whether parent/guardian assessments of their child's recovery correlate with self-reports. At Great Ormond Street a significant proportion of children are unable to answer for themselves. If parent/guardian responses represent a good approximation then this questionnaire may have a role in assessing the quality of recovery in a population of children who are difficult to care for.

DETAILED DESCRIPTION:
In adults a number of instruments have been developed that measure quality of recovery following surgery. The best of these, and the most extensively utilised in other studies, is the QoR-40 (quality of recovery questionnaire with 40 items) developed by Myles and colleagues. QoR-40 is a global measure of recovery incorporating five dimensions; patient support, comfort, emotions, physical independence and pain. They developed this questionnaire from their database of 10,000 patients who had been contemporaneously interviewed about their postoperative experiences. A recent meta-analysis found QoR-40 to be a high-quality instrument, sensitive to clinical change and appropriate for purpose.

The only significant problem with QoR-40 is the time taken to complete it; an average of just over 6 minutes. In response to this the same group developed a shorter version, QoR-15 (quality of recovery questionnaire with 15 items) incorporating elements from all five original domains. The QoR-15 has been validated in adults and correlates well with QoR-40 and takes only 2.5 minutes to complete. However, the average age of the test population was 56 years (+/- 16 years) with a range from 18 to 85 years.

QoR-15 has not been used previously in children, so in preparation for this study the investigators trialed it in ten children to assess its basic acceptability. The investigators also carried out more extensive cognitive interviews in 5 children to assess whether children interpreted the meaning of the questions as intended. As a consequence, minor modifications have been made to the wording of some questions. For example, a question about feeling able to return to work has been changed to a question about feeling able to return to school/ college. The investigators also changed a question asking about the presence of moderate pain to a question about any pain, as children did not distinguish between moderate and mild pain and interpreted the original question as meaning low levels or any pain.

The visual representation of the scoring scheme has also been modified, as children found the original QoR-15 scales confusing. This will not affect the final scoring or the weighting given to any question in any way, it simply makes the scoring easier for children to understand. This modified questionnaire has been termed the PaedQoR-15 and it is this version that will be assessed in our patient population.

ELIGIBILITY:
Inclusion Criteria:

* Child/ young person undergoing general anaesthesia for surgery or diagnostic imaging

Exclusion Criteria:

* English language skills of either parent/guardian or child inadequate to allow informed consent and/or comprehension of the questionnaire
* Intellectual disability precluding adequate comprehension of the questionnaire
* Clinical condition of child precluding adequate comprehension of the questionnaire e.g. preoperative ventilation, reduced level of consciousness
* Emergency admissions where there is insufficient time to allow informed consent

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children/ young people aged between 10 and 18 years undergoing general anaesthesia for surgery or diagnostic imaging
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in PaedQoR-15 between preoperative and one-day postoperative scores | 24 hours

SECONDARY OUTCOMES:
Efficacy of PaedQoR-15; measured by validity, reliability, responsiveness and acceptability | 24 hours
  Psychometric evaluation of modified questionnaire in this new patient population
Parental responses | 24 hours
  Correlation of child/ young person with parent/ guardian scores

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Rawlinson, FRCA MA, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust